CLINICAL TRIAL: NCT06867939
Title: A Pilot Study of Curcumin (Soloways ™) in Patients With Inflammatory Bowel Disease Homozygous for the IL-10 Variant
Brief Title: A Study of Curcumin (Soloways ™) in Patients With Inflammatory Bowel Disease Homozygous for the IL-10 Variant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: S.LAB (SOLOWAYS) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SW019
Record Dates: First submitted 2025-02-20; First posted 2025-03-10 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-03

CONDITIONS: Inflamatory Bowel Disease
Keywords: inflamatory bowel; inflammation; Interleukins; IL-10; supplements; curcumin
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IL-10 Homozygous Variant Cohort (Experimental)
  Interventions: Dietary Supplement: liposomal curcumin
- Non-Variant (Control) Cohort (Active Comparator)
  Interventions: Dietary Supplement: Liposomal Curcumin

INTERVENTIONS:
Dietary Supplement: liposomal curcumin — Liposomal Curcumin, 400-600 mg/day taken orally for 12 weeks, plus standard of care.
  Arms: IL-10 Homozygous Variant Cohort
Dietary Supplement: Liposomal Curcumin — Liposomal Curcumin, 400-600 mg/day taken orally for 12 weeks, plus standard of care.
  Arms: Non-Variant (Control) Cohort

SUMMARY:
This pilot, genotype-stratified clinical trial aims to evaluate the safety and preliminary efficacy of liposomal curcumin in patients with inflammatory bowel disease (IBD) who are homozygous for a specific "unfavorable" IL-10 gene variant (e.g., rs1800896). The study will compare clinical and inflammatory markers in two cohorts: (1) homozygous carriers of the IL-10 variant and (2) non- carriers. The hypothesis is that curcumin supplementation will lead to more pronounced improvement in clinical activity scores and inflammatory biomarkers among homozygous carriers due to their inherently reduced anti-inflammatory capacity.

DETAILED DESCRIPTION:
Inflammatory bowel diseases (including Crohn's disease and ulcerative colitis) are characterized by chronic intestinal inflammation driven by a complex interplay of genetic, immune, and environmental factors. IL-10 plays a crucial role in anti-inflammatory pathways; certain genetic variants can reduce IL-10 production and predispose patients to more severe disease phenotypes.

Curcumin, a polyphenol derived from turmeric, has shown anti-inflammatory effects via multiple molecular targets, including NF-κB. However, curcumin's bioavailability is limited; liposomal formulations may enhance its absorption and therapeutic impact. This pilot trial examines whether liposomal curcumin provides a more significant clinical benefit specifically in patients with the homozygous IL-10 variant, as this subgroup may be particularly responsive to additional anti- inflammatory support.

ELIGIBILITY:
Inclusion Criteria:

- Adults aged 18-70 years with a confirmed diagnosis of ulcerative colitis or Crohn's disease.

Stable background IBD treatment regimen (5-ASA, immunomodulators, or low-dose corticosteroids) for at least 4 weeks prior to enrollment.

* Willingness to undergo genotyping for the IL-10 variant and to comply with the study protocol.
* For the IL-10 Homozygous Variant Cohort: confirmed homozygous "unfavorable" variant (e.g., rs1800896) prior to enrollment. 5. For the Non-Variant Cohort: confirmed absence of the "unfavorable" allele (wild-type).

Exclusion Criteria:

* Use of high-dose corticosteroids or biologics (e.g., TNF inhibitors) initiated within 4 weeks prior to enrollment.
* Known allergy or hypersensitivity to curcumin or related compounds. Severe concomitant illness (significant liver or renal dysfunction, uncontrolled diabetes, etc.) that could interfere with interpretation of results or patient safety.
* Pregnancy or breastfeeding.
* Inability to provide informed consent or comply with study procedures.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-05-05 (Actual); Primary Completion 2024-09-20 (Actual); Study Completion 2025-02-02 (Actual)

PRIMARY OUTCOMES:
Change in Clinical Disease Activity Index | 12 weeks
  Change in the Mayo Clinic Score from baseline to 12 weeks will be assessed for patients with ulcerative colitis. The Mayo Clinic Score is a composite index with four components (stool frequency, rectal bleeding, endoscopic findings, and physician's global assessment), each rated 0 to 3, resulting in a total score ranging from 0 to 12. Higher scores indicate worse disease activity.
For Crohn's disease: Crohn's Disease Activity Index | 12 Weeks
  Change in the Crohn's Disease Activity Index (CDAI) from baseline to 12 weeks will be assessed for patients with Crohn's disease. The CDAI is calculated from multiple clinical variables and typically ranges from 0 to approximately 600, with higher scores indicating more active disease.

SECONDARY OUTCOMES:
Change in High-sensitivity C-Reactive Protein (hs-CRP) Concentration | 12 weeks
  Change in serum high-sensitivity C-reactive protein (hs-CRP) concentration (measured in mg/L) from baseline to 12 weeks. The outcome will be reported as the mean change in hs-CRP concentration.
Change in Fecal Calprotectin Concentration | 12 weeks
  Change in fecal calprotectin concentration (measured in µg/g) from baseline to 12 weeks will be assessed. The outcome will be reported as the mean change in fecal calprotectin concentration.
Change in Additional Cytokines TNF-α | 12 weeks
Change in Additional Cytokines IL-1β | 12 weeks
Adverse Events | 12 weeks
Change in Patient-Reported Quality of Life as Measured by the Inflammatory Bowel Disease Questionnaire (IBDQ) | 12 weeks
  Description: Patient-reported quality of life will be assessed using the Inflammatory Bowel Disease Questionnaire (IBDQ). The IBDQ total score ranges from 32 to 224, where higher scores indicate a better quality of life. The outcome will be reported as the mean change in IBDQ total score from baseline to 12 weeks.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for New Medical Technologies, Novosibirsk, Russia

IPD SHARING:
Plan to Share IPD: No